CLINICAL TRIAL: NCT00901914
Title: A Multi-national, Randomised, DBPC, Phase II Study to Assess the Efficacy and Safety of Three Doses of SLIT Administered as rBet v 1 Tablets Once Daily to Patients Suffering From Birch Pollen Rhinoconjunctivitis
Brief Title: Study of rBet v1 Tablets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Collaborators: Quintiles, Inc. (Industry); Aptuit (Industry)
Responsible Party: Bruno ROBIN, Stallergenes SA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO59.08; 2007-007869-21 (EudraCT Number)
Record Dates: First submitted 2009-04-28; First posted 2009-05-14 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2010-02

CONDITIONS: Birch Pollen-related Rhinoconjunctivitis; Rhinitis, Allergic, Seasonal
Keywords: Hypersensitivity; Allergy; Birch, allergy, Sublingual Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- 2 (Experimental): 12.5 µg rBet v 1
  Interventions: Biological: rBet v 1
- 3 (Experimental): 25 µg rBet v 1
  Interventions: Biological: rBet v 1
- 4 (Experimental): 50 µg rBet v 1
  Interventions: Biological: rBet v 1

INTERVENTIONS:
Biological: Placebo — One sublingual tablet of matching placebo daily during approximately 5.5 months
  Other Names: Placebo control
  Arms: 1
Biological: rBet v 1 — One sublingual tablet containing rBet v 1 at a dosage of 12.5 µg daily during approximately 5.5 months
  Other Names: rBet v 1.0101
  Arms: 2
Biological: rBet v 1 — One sublingual tablet containing rBet v 1 at a dosage of 25 µg daily during approximately 5.5 months
  Other Names: rBet v 1.0101
  Arms: 3
Biological: rBet v 1 — One sublingual tablet containing rBet v 1 at a dosage of 50 µg daily during approximately 5.5 months
  Other Names: rBet v 1.0101
  Arms: 4

SUMMARY:
The purpose of this study is to determine the efficacy and safety of three doses of r Bet v1 administered as sublingual tablets in birch pollen allergic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic birch pollen-related allergic rhinoconjunctivitis for at least the last 2 pollen seasons
* Sensitisation to birch pollen as demonstrated, at screening, by a positive SPT to birch pollen with wheal diameter greater than 3 mm and specific IgE levels > 0.70 kU/L (birch pollen and rBet v 1)
* Patients asymptomatic to all other allergens during the birch pollen season
* RRTSS during the previous pollen season ≥ 12 out of a maximum possible score of 18
* Patients with an FEV1 ≥ 80% of the predicted value
* Female patients with no childbearing potential
* Female patients of childbearing potential are eligible if they are not sexually active or if they use a medically accepted contraceptive method and have a negative urine pregnancy test, and are willing and able to sign written informed consent stating that they will use appropriate contraception and not plan a pregnancy during this study
* Patients able to be compliant with respect to the completion of the daily record card and taking of the investigational products
* Patients having provided signed informed consent

Exclusion Criteria:

* Patients with symptoms of rhinoconjunctivitis during the birch pollen season due to non-birch-related allergens
* Patients with symptomatic allergic rhinitis/rhinoconjunctivitis due to house dust mites
* Patients with symptomatic allergic rhinitis/rhinoconjunctivitis due to cat or dog allergens, and living with these animals at home or at risk of frequent contacts with these animals (family, friends etc.) during the course of the study
* Patients who previously received desensitisation treatment to birch pollen and/or another Betulaceae sp. within the previous 10 years
* Patients with asthma (except birch seasonal asthma in which case the patient could be included in the study)
* Patients with any nasal or oral condition that could interfere with efficacy or safety assessments (such as nasal polyposis or oral inflammation)
* Patients with a past or current disease, which as judged by the investigator, may affect the patient's participation in or outcome of this study
* Any disease or condition which would place a patient at undue risk by being included in the study (according to the investigator's opinion)
* Usual contra-indications of immunotherapy such as concomitant local or systemic beta-blocker therapy and/or immunosuppressive drugs
* Patients with ongoing treatment by immunotherapy with another allergen
* Patients treated with inhaled/systemic steroids within 4 weeks prior to Screening, or with long acting systemic corticosteroids 12 weeks before Screening
* Patients under continuous corticotherapy or undergoing chronic treatment with H2-antihistamine drugs
* Known hypersensitivity to mannitol
* Pregnancy, breast-feeding/lactation or sexually active women of childbearing potential who are not using a medically accepted contraceptive method
* Patients with a history of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Average Adjusted Symptom Score | ~1 month (whole birch pollen season)

SECONDARY OUTCOMES:
Average Rhinoconjunctivitis Total symptom Score | ~1 month (whole birch pollen season)
Rescue Medication Score | ~1 month (whole birch pollen season)
Average Combined Score | ~1 month (whole birch pollen season)
Proportion of symptom-controlled days | ~1 month (whole birch pollen season)
Global evaluation by the patient | after 5-6 months of treatment
Immunological markers (IgE and IgG4) | 6-7 months
Sensitisation status | At least 6 months
Lower airways symptoms | ~1 month (whole birch pollen season)
Safety assessments | 6-7 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Rak, MD. PR, Principal Investigator — Sahlgrenska University Hospital, Department of Respiratory Medicine and Allergy, 413 45 Gothenburg, Sweden
Locations (8):
- National University Hospital - Allergy Unit 4222, Copenhagen, Denmark
- Helsingin yliopistollinen keskussairaala, Helsinki, Finland
- NHC, Hôpitaux Universitaires de Strasbourg, Strasbourg, France
- Charité universitaetsmedizin, Berlin, Germany
- Public Institution Kaunas Medical University Hospital, Kaunas, Lithuania
- SPZOZ Uniwersytecki Szpital Kliniczny Nr 1im.N.Barlickiego w Uniwersystetu Medycznego w Łodzi, Lodz, Poland
- Institute of Immunology of FMBA, Moscow, Russia
- Sabina RAK, Gothenburg, Sweden